CLINICAL TRIAL: NCT06019312
Title: The Impact of Lactobacillus Plantarum 299v in Combination With Inulin on Gut Microbiome, Chemotherapy and Radiotherapy-induced Diarrhoea, and Clostridioides Difficile Infection in Colorectal Cancer Patients in Periooperative Period
Brief Title: L. Plantarum 299v and Gut Microbiome, Diarrhoea, and Clostridioides Difficile Infection in Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUGdansk_Lp299v
Record Dates: First submitted 2023-08-10; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer; Clostridioides Difficile Infection; Diarrhea
Keywords: Lactobacillus plantarum 299v; Probiotics; Colorectal Cancer; Clostridioides difficile; Diarrhea
MeSH Terms: conditions — Colorectal Neoplasms; Clostridium Infections; Diarrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lactobacillus plantarum 299v (Experimental): 15 patients will receive 2 capsules (per day - 1 capsule contains 10x10 CFU) of L. plantarum 299v for 4 weeks
  Interventions: Dietary Supplement: Sanprobi IBS®
- Lactobacillus plantarum 299v in combination with inulin (Experimental): 15 patients will receive 2 capsules (per day - 1 capsule contains 10x10 CFU) of L. plantarum 299v and inulin (4 g) for 4 weeks
  Interventions: Dietary Supplement: Sanprobi IBS®
- Placebo in combination with inulin (No Intervention): 15 patients will receive 2 capsules (per day) of placebo and inulin (4 g) for 4 weeks
- Placebo (No Intervention): 15 patients will receive 2 capsules (per day) of placebo for 4 weeks

INTERVENTIONS:
Dietary Supplement: Sanprobi IBS® — Patients will be treated with probiotics in combination with inulin, which is able to stimulate the growing of probiotic bacteria in gastrointestinal tract.
  Arms: Lactobacillus plantarum 299v; Lactobacillus plantarum 299v in combination with inulin

SUMMARY:
Colorectal cancer in periooperative period patients (n=60) will be enrolled to this study. Participants will be divided into 4 groups as follows:

* group 1 (n=15) will receive 2 capsules (per day) of L. plantarum 299v L. plantarum 299v (Sanprobi IBS®) for 4 weeks
* group 2 (n=15) will receive L. plantarum 299v (2 capsules per day) and inulin (4 g) for 4 weeks
* group 3 (n=15) will receive placebo (2 capsules per day) and inulin (4 g) for 4 weeks
* group 4 (n=15) will receive placebo (2 capsules per day) for 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 oraz ≤65
* patients with colorectal cancer prior to surgical treatment
* qualification to surgery
* the treatment with chemotherapy and radiotherapy in preoperative period
* an appropriate swallowing
* patients agreement to take part in this study

Exclusion Criteria:

* the presence of other cancers than colorectal cancer
* inflammatory bowel diseases
* dysphagia
* intake of antibiotics, proton pump inhibitors, probiotics, and synbiotics 3 months befor taking part in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
gut microbiota composition | 4 weeks
  It will be measured by presenting alpha diversity and beta-diversity of microbial community and after that it will be presented using bioinformatic analysis.

SECONDARY OUTCOMES:
chemotherapy and radiotherapy-induced diarrhoea | 4 weeks
  It will be analysed by using own created survey.
Clostridioides difficile infection | 6 months
  The incidence of Clostridioides difficile infection will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Surgery with Unit of Oncological Surgery in Koscierzyna, Kościerzyna, Poland

IPD SHARING:
Plan to Share IPD: Undecided